CLINICAL TRIAL: NCT05618392
Title: Pain Assessment Following Placement of a Percutaneous Radiologic Gastrostomy and Predictive Factors
Acronym: DOULEURGPR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Valence (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH-CHV-11
Record Dates: First submitted 2022-06-03; First posted 2022-11-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Gastrostomy Complications; Gastrostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group assignment: only one arm. Each patient complete numerical scale questionnaire (0-10)

SUMMARY:
A 12 months mono-center, descriptive study, to evaluate pain and predictive factors Following placement of percutaneous Radiologic gastrostomy (PRG).

The primary objective is to evaluate the abdominal pain associated with percutaneous radiologic gastrostomy (PRG) placement.

DETAILED DESCRIPTION:
PRG is a pathway first of all enteral nutrition that has several advantages: local anesthesia, possible in case of esophageal stenosis, Rates of successful tube placement higher for radiologic gastrostomy than for percutaneous endoscopic Gastrostomy (PEG).

Abdominal pain following percutaneous radiologic gastrostomy (PRG) placement is a recognized complication. However, the prevalence and degree of severity of pain are poorly characterized. This pain often requires antalgic treatment.

The primary objective is to evaluate the abdominal pain from Baseline until 7 days after radiologic gastrostomy (PRG) placement.

The secondary objective is to evaluate predictive factors

ELIGIBILITY:
Inclusion Criteria:

* Needing a radiologic gastrostomy under local anesthesia
* Age ≥ 18 years old
* Read, write and understand the French language

Exclusion Criteria:

* Patient under guardianship, deprived of liberty, safeguard of justice
* Patient presenting a serious psychiatric pathology that does not allow compliance with the completion of the questionnaires (at the discretion of the investigator)
* Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients needing a Percutaneous radiologic Gastrostomy under local anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
abdominal pain | 7 days
  numerical scale 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
predictive factors | DAY 1
  determine predictive factors of pain suspected in advance:
  * Fasting anterior stomach wall depth estimated during the ultrasound survey(mm)
  * Gastric topography determined under X-ray (subcostal / partially retrohepatic)
  * Topography of the anchors: large tuberosity / antrum
  * Distance of anchors from each other (mm)
  * Depth of the anchors (mm)
  * Skin depression of anchors: (with depression, without depression)
  * Intraparietal length of the gastrostomy tube (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Sandrine Beauchard, Valence, France

IPD SHARING:
Plan to Share IPD: Undecided